CLINICAL TRIAL: NCT00099216
Title: Efficacy and Safety of Rivastigmine Capsules in Patients With Probable Vascular Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CENA713BIA05
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Vascular Dementia
Keywords: Dementia,vascular,rivastigmine,stroke,memory loss
MeSH Terms: conditions — Dementia, Vascular; Dementia | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine

SUMMARY:
The goal of this research study is to evaluate the effectiveness, tolerability and safety of rivastigmine capsules in males and females between the ages of 50 and 85 years old with probable vascular dementia.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50 and 85 years old
* Have contact with a responsible caregiver 3 or more days per week
* Be male or a female who is surgically sterilized or one year post menopausal

Exclusion Criteria:

* Current diagnosis of severe or unstable cardiovascular or other diseases
* Current diagnosis of active, uncontrolled seizure disorder, Parkinson's disease or Alzheimer's disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2001-08; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change in cognition from baseline at week 24
Global clinical impression of change from baseline at week 24

SECONDARY OUTCOMES:
Change in activities of daily living from baseline at week 24
Change in behavioral symptoms from baseline at week 24
Change in clinical staging from baseline at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (63):
- United States (17):
  - Irvine, California
  - San Francisco, California
  - Boynton Beach, Florida
  - Miami Beach, Florida
  - Port Charlotte, Florida
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Greensburg, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Houston, Texas
  - Bennington, Vermont
- Austria (3):
  - Graz
  - Linz
  - Vienna
- Canada (4):
  - Edmonton, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (7):
  - Amiens
  - Bordeaux
  - Lille
  - Marseille
  - Montpellier
  - Toulouse
  - Tours
- Germany (9):
  - Bautzen
  - Berlin
  - Bochum
  - Chemnitz
  - Eisenhüttenstadt
  - Erlangen
  - Freiburg im Breisgau
  - Lüdenscheid
  - Osnabrück
- Italy (7):
  - Ancona
  - Brescia
  - Florence
  - Perugia
  - Reggio Emilia
  - Roma
  - Vicenza
- Russia (2):
  - Moscow
  - Saint Petersburg
- Spain (5):
  - Barakaldo
  - Barcelona
  - Madrid
  - Pamplona
  - Saint Cugat Del Valles
- Switzerland (2):
  - Basel
  - Lausanne
- United Kingdom (7):
  - Newcastle upon Tyne, Newcastle
  - Swindon, Wiltshire
  - Bristol
  - Clydebank
  - East Sussex
  - Lytham St Annes
  - Southampton

REFERENCES:
- [Derived] Ballard C, Sauter M, Scheltens P, He Y, Barkhof F, van Straaten EC, van der Flier WM, Hsu C, Wu S, Lane R. Efficacy, safety and tolerability of rivastigmine capsules in patients with probable vascular dementia: the VantagE study. Curr Med Res Opin. 2008 Sep;24(9):2561-74. doi: 10.1185/03007990802328142. Epub 2008 Jul 31. PMID 18674411
- See also: Click here for further information and to find an investigational site near you — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=331&diseaseID=31zip=07430